CLINICAL TRIAL: NCT05542745
Title: Rate of Upper Incisors Retraction in Class II Division 1 Patients Managed With Palatal Versus Buccal Miniscrew Supported Segmental Orthodontics: Randomized Clinical Trial
Brief Title: Measuring Rate of Anteriors Retraction With Two Different Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10061119
Record Dates: First submitted 2022-09-11; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Orthodontics, incisors retraction, mini-implants, direct- anchorage.
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palatal retractor (Active Comparator): palatal retraction
  Interventions: Device: palatal and buccal retraction
- buccal retractor (Active Comparator): buccal retraction
  Interventions: Device: palatal and buccal retraction

INTERVENTIONS:
Device: palatal and buccal retraction — comparison

SUMMARY:
Few studies had investigated the effectiveness of segmental retraction. As a result of that, this study was concerned about comparing retraction rate of maxillary incisors between buccal and palatal mini-implant supported retraction groups in Class II division 1 non growing patients for 3 months interval.

DETAILED DESCRIPTION:
Almost all patients their primary concern is the total duration of orthodontic treatment. So, the need to choose the best mean to fasten the tooth movement rate with least drawbacks increased . Many new bracket techniques and prescriptions have been evolved since straight wire technique of Andrew's was advanced. All of these progressions are to make a system of force which can decrease the overall management time.

Commonly, extractions and maximum anchorage are planned to manage different malocclusions in orthodontic treatment especially in protrusion cases. Space closure is an important step following extraction. So, space closure strategy must be individually adjusted depending on diagnosis and plan of treatment. Nowadays several options are used to fasten movement of tooth. New techniques like implants assisted retraction, lessen the time of retraction and accordingly the total time of treatment.

Control of anchorage is an important factor in orthodontic therapy success. Mini-implants are method of absolute anchorage control .These systems improves the anchorage, but still have some drawbacks like surgical intervention and patient compliance. However, their usage becomes a necessity and unavoidable in many cases. Buccal TADs could provide superior results when retracting anterior teeth in patients with moderate to severe protrusion.

Lingual orthodontics introduction created novel horizons in orthodontic therapy. Labial orthodontics varied differentially in biomechanics from the lingual one. Because of its positional biomechanical advantage, lingual orthodontics offers higher anchorage and higher rate of retraction; as the lingual appliance force applied near to the tooth center of resistance than in the labial ones.

Control of torque is not simple in traditional lingual orthodontics. The C-lingual retractor is great for lip protrusion cases that need maximum anchorage.Bonding the C-retractor to the palatal aspect of the upper anteriors, adding maximum esthetics. Mini-implants are inserted palataly and decrease the need of posterior anchorage for retraction of upper anterior teeth. This is named lingual biocreative therapy. Palatal TSADs can provide wide range of force application level, due to the depth of palatal vault. By the adjustment of the lever arm length and position of miniscrews, the desired line of action of the retraction force with respect to the center of resistance of the anterior segment can be achieved.Segmental retraction is an approach using palatal TSADs as direct anchorage. The anterior teeth were splinted on the lingual side, and they are retracted to the palatal TSADs using elastomers or NiTi coil springs through a lever connected to the anterior segment.

It is critical to locate and manage the center of resistance relative to the force vector of retraction. By using this, the orthodontist can estimate the power arm length which would provide controlled tipping, or bodily movement of the anterior area.

There is a lack of studies evaluating the rate of movement of incisors in cases treated with palatal retraction so new investigations are needed in this area. Because of the biomechanical differences between buccal and palatal retraction, this study targeted the comparison of the rate of retraction in upper anteriors following leveling and alignment in class II division 1 patients managed by either method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Class II division 1 malocclusion with no or mild crowding 2. Age ranging from 14 to 18 years.

Exclusion Criteria:

* No previous orthodontic therapy of any type prior to this treatment No systematic disease Good oral hygiene and no periodontal problems No abnormal oral habits

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
rate of retraction | 3 months
  distance travelled at specific time interval

CONTACTS AND LOCATIONS:
Overall Officials: ElBialy, Principal Investigator — Faculty of Dentistry Mansoura Univesity
Locations (1):
- Egypt, Al Mansurah, Egypt